CLINICAL TRIAL: NCT03750682
Title: ENhancing Independence Using Group-Based Community Interventions for Healthy AGing Elders: The ENGAGE for Brain Health Pilot Study
Brief Title: ENGAGE for Brain Health
Acronym: ENGAGE-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Boston Older Americans Independence Center (Unknown); Somerville Council on Aging, Massachusetts (Unknown)
Responsible Party: Principal Investigator, Kieran Reid, Scientist II, Tufts University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13136
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Motoric Cognitive Risk Syndrome
MeSH Terms: interventions — Exercise; Methods; Helium

STUDY DESIGN:
Intervention Model Description: The ENGAGE for Brain Health is designed as a single blind, randomized-controlled, parallel group pilot study. This study plans to enroll up to 40 participants to be randomized into the PA or HE intervention group.
Masking Description: No one is blinded during this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention (PA) (Active Comparator): The PA intervention will consist of a twice per week group-based moderate-intensity program that includes aerobic, strength, flexibility, and balance training.
  Interventions: Other: Physical Activity (PA) Intervention
- Health Education Intervention (HE) (Placebo Comparator): The HE intervention will consist of bimonthly lifestyle counseling workshops in a group setting. Participants will receive information on a variety of topics including relevance to older adults, including nutrition, understanding the health care system, dietary guidelines for older adults, safe travel, age-appropriate preventive services, information on resources, etc.
  Interventions: Other: Healthy Aging Education (HE) Intervention

INTERVENTIONS:
Other: Physical Activity (PA) Intervention — The PA intervention will consist of a twice per week group- based moderate-intensity multimodal program that includes aerobic, strength, flexibility, and balance training, as previously described. The Community Health Promoter will be trained and certified by Dr. Reid to deliver the PA intervention. PA will be conducted at the Holland Street Senior Center in Somerville, MA. The center is equipped with a large dining hall and corridors which will be utilized to perform the various components of the PA intervention for ENGAGE-B. This real-world approach was shown to be safe, feasible and effective in the initial ENGAGE study among older adults with severe mobility-limitations. Throughout PA, walking will be the primary mode of exercise, given its widespread applicabilityThe study staff will administer an Adverse Event/Concomitant Medication Questionnaire biweekly to all PA subjects.
  Arms: Physical Activity Intervention (PA)
Other: Healthy Aging Education (HE) Intervention — The HE intervention will also be conducted at the Holland Street Senior Center in Somerville, MA. Participants will receive bimonthly lifestyle counseling workshops in a group setting. Participants will receive information on a variety of topics of relevance to older adults (e.g., nutrition for brain health, effective negotiation of the health care system, dietary guidelines for older adults, safe travel, age-appropriate preventive services and screenings, resources for reliable health information, etc.). All intervention materials will be submitted for IRB approval prior to the presentation. In addition to educational offerings, an instructor led program (5-10 minutes) of gentle upper extremity stretching exercises and relaxation techniques are to be performed during each class.
  The study staff will administer an Adverse Event/Concomitant Medication Questionnaire biweekly to all HE subjects.
  Arms: Health Education Intervention (HE)

SUMMARY:
Age-related cognitive decline has a profound impact on the daily functioning of older adults, their families and healthcare systems. Despite its significant personal, societal and economic impact, no pharmacologic therapies presently exist to mitigate age-related cognitive decline. As the population of older adults continues to rapidly increase, the implementation of effective and scalable low-cost interventions that may maintain the cognitive independence of broad populations of older persons are now of urgent public health priority.

DETAILED DESCRIPTION:
ENGAGE-B is a single blind, parallel-group, community-based randomized controlled pilot study. The overall objective of the study is to build on our recently completed ENGAGE pilot study and further examine and characterize the feasibility and effectiveness of translating the LIFE study physical activity intervention (PA) into a real-world community-based senior center setting. ENGAGE-B will target the recruitment of older adults with subjective memory complaints and slow gait (motoric cognitive risk syndrome (MCR)). Participants with MCR will be randomized to a 24-week PA intervention (n = 20) or to a healthy aging education control intervention (HE) (n = 20). ENGAGE-B will also test a highly practical and scalable innovation for the delivery of exercise programming for at-risk older adults in the community setting. An existing community-based senior center employee ("Community Health Promoter"), without a formal background in exercise physiology, will be trained by the study investigators to deliver the PA intervention among older adults with MCR. The primary feasibility outcomes will be assessed by quantifying intervention adherence and the occurrence of adverse events across the PA and HE intervention arms. Secondary and exploratory outcomes will include the comparative evaluation of specific domains of cognitive performance (executive function, global cognition, working memory, computerized cognitive testing and complex walking tasks), non-invasive functional near-infrared spectroscopy (fNIRS) derived measures of prefrontal brain activation, mobility, accelerometry-derived estimates of physical activity, depression, quality of life and costs associated with delivering the respective interventions. Results from this proposed pilot study are intended as the basis for a larger and more definitive pragmatic trial in older adults. If successful this pilot work will serve as an exciting preliminary model to potentially target and mitigate the loss of cognitive independence across a variety of community-based locations.

ELIGIBILITY:
Inclusion Criteria:

* • Men and Women age 60-89 years, community-dwelling, ambulatory

  * Presence of MCR syndrome
  * Sedentary (reporting ≤ 20 min/week of regularly structured physical activity in the past month)
  * Written permission from PCP for study participation
  * Willingness to be randomized and participate for 24 weeks

Exclusion Criteria:

* • Acute or terminal illness

  * Modified Mini-Mental State Examination Score <80(<76 if African American)*
  * Myocardial Infarction in the previous 6 months
  * Symptomatic coronary artery disease
  * Upper or lower extremity fracture in the previous 6 months
  * Resting blood pressure >180/100 mmHg
  * Unable to communicate due to severe hearing loss or speech disorder
  * Severe visual impairment that may preclude participation in the study assessments or interventions
  * Non-English speaking

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Measuring the safety of a 6 month PA or HE intervention in a community setting in older adults with MCR | 6 Months
  Safety will be measured by the number of adverse events and serious adverse events. The investigators will compare the rates of adverse events and serious adverse events between the physical activity and healthy aging education intervention randomized arms.
Measuring the success (feasibility) of integrating clinical exercise programs into real-world community-based settings. | 6 Months
  Feasibility will be measured by adherence to PA by percent attendance. Successful adherence will be defined by an attendance rate of >60%.

SECONDARY OUTCOMES:
fNIRS (Functional Near-Infrared Spectroscopy) assessment and submaximal cycle ergometry | 6 Months
  We will utilize Functional Near-Infrared Spectroscopy (fNIRS) to non-invasively evaluate the brain hemodynamics of participants during a single bout of moderate intensity submaximal cycling exercise.
Accelerometry | 6 Months
  Regular activity level will be measured using accelerometry (GT3X+, Actigraph, Pensacola, FL). The actigraph, attached to an elastic belt, will be worn around the waist of the participant. These accelerometers are small enough to be unobtrusive and produce little interference with normal physical activity. Participants will be instructed to wear the actigraph for a 7-day period during waking hours and remove it for sleep and bathing only. Activity will be recorded using 1-second epochs.
6-Minute Walk Test (6MWT) | 6 Months
  The 6MWT tests functional exercise capacity by measuring the distance a participant can walk within a 6 minute time period. The 6MWT is a beneficial tool in assessing functional exercise capacity in older adults. The 6MWT will be performed in a corridor of the Holland Street Senior Center in Somerville, MA on a 40 meter course. Participants will be instructed to walk as far as they can in six minutes without running or jogging. Cones will be set up at each turnaround point of the course and participants will be instructed to complete as many laps as they can without overexerting themselves. The test will be stopped if any of the following symptoms occur: chest pain, severe dyspnea, muscle cramping, diaphoresis, or any other symptom the investigator deems unsafe. Subjects' walking distance will be recorded.
Grip Strength Test | 6 Months
  Hand grip strength will be measured in the dominant hand with a Jamar Handheld Dynamometer (Patterson Medical, Warrenville, IL). The participants will perform the test while sitting comfortably with shoulder adducted and neutrally rotated, the elbow supported on a table and flexed to 90 degrees, forearm and wrist in neutral position. The patients will be instructed to perform a maximal isometric contraction. The test will be repeated after 10 sec. and the highest value will be recorded.
Complex Walking Tasks (CWT's) | 6 Months
  During the CWTs, subjects will first be asked to walk on an even surface for 7 meters, as fast as possible while remaining safe. Subjects will be then asked to repeat the walk in their usual pace at the same time as subtracting 3 from 50 and keep subtracting until the 7 meters walk is completed. Subjects' complex walking speed will be timed with a stopwatch and each subtraction will be recorded.
Quality of Well Being | 6 Months
  The self-administered version of the Quality of Well-Being Scale will be used to assess general quality of life. This instrument provides a comprehensive measure of health-related quality of life that assesses health symptoms and functioning. This scale has 6 parts. Part 1: acute and chronic symptoms, part 2: self care, part 3: mobility, part 4: physical activity, part 5: usual activity, part 6: general health. There are 79 questions total. Each question is uses the scale: have you... in the past 0 days, 1 day, 2 days, 3 days. There is no scoring or total scoring mechanism. Outcome depends on the question being asked. For example, if a participant reports no hospital visits in the past 3 days that is considered better than reporting no hospital visits in the past 1 day.
Falls Efficacy Scale-International | 6 Months
  The Falls Efficacy Scale-International is a questionnaire that evaluates the fear of falling among community dwelling older adults. This questionnaire will be administered at baseline and 24 weeks.
Fall History | 6 Months
  Participants will be asked about any recent falls they have experienced at each assessment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kieran Reid, PhD, MPH, Principal Investigator — Jean Mayer Human Nutrition Research Center on Aging at Tufts University
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid KF, Laussen J, Bhatia K, Englund DA, Kirn DR, Price LL, Manini TM, Liu CK, Kowaleski C, Fielding RA. Translating the Lifestyle Interventions and Independence for Elders Clinical Trial to Older Adults in a Real-World Community-Based Setting. J Gerontol A Biol Sci Med Sci. 2019 May 16;74(6):924-928. doi: 10.1093/gerona/gly152. PMID 30010808
- [Background] Wimo A, Guerchet M, Ali GC, Wu YT, Prina AM, Winblad B, Jonsson L, Liu Z, Prince M. The worldwide costs of dementia 2015 and comparisons with 2010. Alzheimers Dement. 2017 Jan;13(1):1-7. doi: 10.1016/j.jalz.2016.07.150. Epub 2016 Aug 29. PMID 27583652
- [Background] Brasure M, Desai P, Davila H, Nelson VA, Calvert C, Jutkowitz E, Butler M, Fink HA, Ratner E, Hemmy LS, McCarten JR, Barclay TR, Kane RL. Physical Activity Interventions in Preventing Cognitive Decline and Alzheimer-Type Dementia: A Systematic Review. Ann Intern Med. 2018 Jan 2;168(1):30-38. doi: 10.7326/M17-1528. Epub 2017 Dec 19. PMID 29255839
- [Background] Gates N, Fiatarone Singh MA, Sachdev PS, Valenzuela M. The effect of exercise training on cognitive function in older adults with mild cognitive impairment: a meta-analysis of randomized controlled trials. Am J Geriatr Psychiatry. 2013 Nov;21(11):1086-97. doi: 10.1016/j.jagp.2013.02.018. Epub 2013 Jul 3. PMID 23831175
- [Background] Allali G, Ayers EI, Verghese J. Motoric Cognitive Risk Syndrome Subtypes and Cognitive Profiles. J Gerontol A Biol Sci Med Sci. 2016 Mar;71(3):378-84. doi: 10.1093/gerona/glv092. Epub 2015 Aug 6. PMID 26248559
- [Background] Verghese J, Wang C, Lipton RB, Holtzer R. Motoric cognitive risk syndrome and the risk of dementia. J Gerontol A Biol Sci Med Sci. 2013 Apr;68(4):412-8. doi: 10.1093/gerona/gls191. Epub 2012 Sep 17. PMID 22987797
- [Background] Rosano C, Chang YF, Kuller LH, Guralnik JM, Studenski SA, Aizenstein HJ, Gianaros PJ, Lopez OL, Longstreth WT Jr, Newman AB. Long-term survival in adults 65 years and older with white matter hyperintensity: association with performance on the digit symbol substitution test. Psychosom Med. 2013 Sep;75(7):624-31. doi: 10.1097/PSY.0b013e31829c1df2. Epub 2013 Jul 25. PMID 23886735
- [Background] Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, Espeland MA, Fielding RA, Gill TM, Groessl EJ, King AC, Kritchevsky SB, Manini TM, McDermott MM, Miller ME, Newman AB, Rejeski WJ, Sink KM, Williamson JD; LIFE study investigators. Effect of structured physical activity on prevention of major mobility disability in older adults: the LIFE study randomized clinical trial. JAMA. 2014 Jun 18;311(23):2387-96. doi: 10.1001/jama.2014.5616. PMID 24866862
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759